CLINICAL TRIAL: NCT05217472
Title: A Phase 2a, Double-Blind, Randomized, Placebo-Controlled Study of Ravagalimab in Subjects With Moderately to Severely Active Primary Sjogren's Syndrome
Brief Title: An Efficacy and Safety Study of Injectable Ravagalimab to Assess Change in EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) in Adult Participants With Moderately to Severely Active Primary Sjogren's Syndrome (pSS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study canceled
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M21-263; 2019-003131-31 (EudraCT Number)
Record Dates: First submitted 2020-02-06; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2020-02

CONDITIONS: Sjogren's Syndrome (SS)
Keywords: Sjogren's Syndrome (SS); Primary Sjogren's Syndrome (pSS); Ravagalimab; ABBV-323
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ravagalimab (Experimental): Participants will receive a loading dose of intravenous (IV) ravagalimab dose A at Week 0 followed by subcutaneous (SC) ravagalimab dose A every other week (eow)
  Interventions: Drug: Ravaglimab; Drug: Ravagalimab
- Placebo (Placebo Comparator): Participants will receive a loading dose of intravenous (IV) placebo at Week 0 followed by subcutaneous (SC) placebo every other week (eow)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ravaglimab — Intravenous Injection
  Other Names: ABBV-323
  Arms: Ravagalimab
Drug: Ravagalimab — Subcutaneous Injection
  Other Names: ABBV-323
  Arms: Ravagalimab
Drug: Placebo — Intravenous Injection
  Arms: Placebo
Drug: Placebo — Subcutaneous Injection
  Arms: Placebo

SUMMARY:
Sjogren's syndrome (SS) is a chronic, multisystem autoimmune disease characterized by lacrimal and salivary gland inflammation, with resultant dryness of the eyes and mouth and occasional glandular enlargement. In addition, a variety of systemic manifestations may occur; including fatigue, musculoskeletal symptoms, rashes, and internal organ (e.g., pulmonary, renal, hepatic, and neurologic) disease. Sjogren's syndrome may occur in isolation, primary Sjogren's syndrome (pSS), or in a secondary form, often associated with rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), or systemic sclerosis. Ravagalimab is an investigational drug being developed to help treat patients with inflammatory diseases like SS. This study will evaluate how well ravagalimab works within the body and how safe it is in patients with primary SS (pSS).

Ravagalimab, a potent CD40 antagonist is an investigational drug being developed for the treatment of Sjogren's syndrome (SS). This study is "double-blinded", which means that neither the trial participants nor the study doctors will know who will be given which study drug. Study doctors put the participants in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to placebo. Participants 18-75 years of age with Sjogren's syndrome (SS) will be enrolled. Around 45 participants will be enrolled in the study in multiple sites within Netherlands.

Participants will receive ravagalimab intravenous (IV) loading dose or IV placebo at baseline followed by subcutaneous (SC) ravagalimab or matching placebo for 22 weeks.

There will be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, labial gland (lip) biopsy, and checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Primary Sjogren's syndrome (pSS) diagnosed according to the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2016 Criteria.
* Lymphocyte focus score (local lymphocytic infiltrates) >= 1 in sublabial salivary gland specimen. Subjects with sublabial salivary gland biopsy obtained 3 months prior to Screening and meeting this criterion will be eligible without a biopsy at Screening. Subjects without a sublabial salivary gland biopsy within 3 months of Screening will obtain a biopsy for a lymphocyte focus score at Screening.
* EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) >= 5 at Screening.
* EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) >= 6 at Screening.

Exclusion Criteria:

* History of clinically significant drug or alcohol abuse within the last 6 months.
* History of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients), the ingredients of Chinese hamster ovary cells and/or other products in the same class.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-06 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) | Week 24
  ESSDAI is a systemic disease activity index including 12 domains (i.e., organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system, central nervous system, haematological, glandular, constitutional, lymphadenopathic and biological).

SECONDARY OUTCOMES:
Change From Baseline in EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) | Up to Week 16
  ESSDAI is a systemic disease activity index including 12 domains (i.e., organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system, central nervous system, haematological, glandular, constitutional, lymphadenopathic and biological).
Change From Baseline in EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | Up to Week 24
  ESSPRI is designed to evaluate the patient symptoms with 3 questions related to the dryness, pain and fatigue a participant has experienced in the prior 2 weeks. It is a numeric rating scale from 0 - 10, with a final score the mean of the 3 questions
Change From Baseline in Tender Joint Count | Up to Week 24
  An assessment of 68 joints will be done for tenderness by pressure manipulation on physical examination. Joint pain/tenderness will be classified as: present, absent, replaced or no assessment.
Change From Baseline in Swollen Joint Count | Up to Week 24
  An assessment of 66 joints will be done by directed physical examination. The joints to be examined for swelling are the same as those examined for tenderness, except the hip joints are excluded. Joint swelling will be classified as present, absent, replaced or no assessment.
Change From Baseline in Salivary Flow (Unstimulated) | Up to Week 24
  Patients will be asked to collect their saliva in a cup every 30 seconds for a total period of 5 minutes. The saliva production is expressed in ml/minute.
Change From Baseline in Salivary Flow (Stimulated) | Up to Week 24
  Saliva production is stimulated by parafilm and collected in a cup every 30 seconds for a total period of 5 minutes.. The saliva production is expressed in ml/minute.
Change From Baseline in Lacrimal Flow (Schirmer's Test of Ocular Function) | Up to Week 24
  Lachrymal flow will be assessed by Schirmer's test of ocular function. A small filter paper will be placed in the conjunctival sac for 5 minutes. After that, the degree of wetting is evaluated
Change From Baseline in Van Bijsterveld Score | Up to Week 24
  The van Bijsterveld score is an ocular score for dryness. The Bijsterveld score is determined by adding up the combined score (from 0 to 3; 0 is normal and 3 is the highest level of staining) in the central and two outer sections of the eye.
Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | Up to Week 24
  FACIT-Fatigue is a 13-item questionnaire that evaluates fatigue/tiredness and its impact on daily activities and functioning in chronic diseases. This instrument includes items such as tiredness, weakness, listlessness, lack of energy, and the impact of these feelings on daily functioning (e.g., sleeping, and social activities). A lower score indicates less negative impact on daily activities.
Change From Baseline in Patient's Global Assessment of Disease Activity Numeric Rating Scales | Up to Week 24
  Patient's Global Assessment of Disease Activity Numeric Rating Scale allows a patient to score 0 - 10 to assess the patient's overall functionality assessment considering the disease activity within the past week
Change From Baseline in Physician's Global Assessment of Disease Activity Numeric Rating Scales | Up to Week 24
  Physician's Global Assessment of Disease Activity Numeric Rating Scale allows a physician to score 0 - 10 to assess the patient's overall functionality assessment considering the disease activity within the past week.
Change from Baseline in anti-Sjogrens-syndrome-related antigen A (anti-SSA) | Up to Week 24
  Change from baseline in anti-SSA s assessed.
Change from Baseline in anti-Sjogrens-syndrome-related antigen B (anti-SSB) | Up to Week 24
  Change from baseline in anti-SSB is assessed.
Change from Baseline in antinuclear antibody (ANA) | Up to Week 24
  Change from baseline in antinuclear antibody (ANA) is assessed.
Change from Baseline in rheumatoid factor (RF) | Up to Week 24
  Change from baseline in rheumatoid factor (RF) is assessed.
Change from Baseline in high-sensitivity C-reactive protein (hsCRP) | Up to Week 24
  Change from baseline in high-sensitivity C-reactive protein (hsCRP) is assessed.
Change from Baseline in immunoglobulin M (IgM) | Up to Week 24
  Change from baseline in immunoglobulin M (IgM) is assessed
Change from Baseline in immunoglobulin M (IgG) | Up to Week 24
  Change from baseline in immunoglobulin M (IgG) is assessed.
Change from Baseline in immunoglobulin A (IgA) | Up to Week 24
  Change from baseline in immunoglobulin A (IgA) is assessed.
Change from Baseline in Serum-Free Light Chains | Up to Week 24
  Change from baseline in serum-free light chains is assessed.
Change from Baseline in Serum C3 | Up to Week 24
  Change from baseline in Serum C3 is assessed.
Change from Baseline in Serum C4 | Up to Week 24
  Change from baseline in Serum C4 is assessed.
Change from Baseline in Haemolytic Complement CH50 | Up to Week 24
  Change from baseline in CH50 is assessed.
Change From Baseline in Focus Score of Sublabial Salivary Gland Biopsy (In Participants With a Screening and Week 24 Biopsy) | Week 24
  Change from baseline in focus score of sublabial salivary gland biopsy is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (1):
- Universitair Medisch Centrum Utrecht /ID# 214029, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html